CLINICAL TRIAL: NCT03198364
Title: Development of a Mobile Heath Augmented Brief Suicide Prevention Intervention for People With SMI Accessing Community Care
Brief Title: Development of a Mobile Heath Augmented Brief Suicide Prevention Intervention for People With SMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Colin Depp, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R34MH113613-01 (NIH); 9370600 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2017-06-20; First posted 2017-06-26 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia; Bipolar Disorder; Suicide and Self-harm
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Suicide; Self-Injurious Behavior | interventions — Safety

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- START + Mobile Augmentation (Experimental): 4 Sessions of In-Person Psychoeducation called Safety and Recovery Therapy (START) with 12 weeks of augmentation by use of automated software to prompt users to engage in personalized adaptive coping
  Interventions: Behavioral: Safety and Recovery Therapy; Behavioral: Mobile Augmentation
- START (Active Comparator): 4 Sessions of In-Person Psychoeducation called Safety and Recovery Therapy (START)
  Interventions: Behavioral: Safety and Recovery Therapy

INTERVENTIONS:
Behavioral: Safety and Recovery Therapy — 4 session individualized psychoeducation tailored to people with bipolar disorder or schizophrenia targeting coping skills for suicidal thoughts and their determinants.
Behavioral: Mobile Augmentation — Though a smartphone device, participants receive 12 weeks of personalized prompts derived from content produced in individual START sessions to increase transfer of skills to day to day life
  Arms: START + Mobile Augmentation

SUMMARY:
Schizophrenia and bipolar disorder are associated with high risk for suicide, yet there are few brief interventions that directly target suicide prevention in this large population. The goal of this intervention development study is to evaluate the feasibility, acceptability, and preliminary effectiveness of a brief intervention called SafeTy and Recovery Therapy (START) that is augmented with content delivered on mobile devices outside of the clinic setting. The intervention will evaluated in a community urgent care center context as people initiate outpatient care, and, if effective, could be deployed in a wide network of such centers.

DETAILED DESCRIPTION:
This intervention development research project evaluates the feasibility, acceptability, and preliminary impact of a brief cognitive behavioral intervention, tailored to SMI, that is delivered during the gap period between urgent care evaluation and follow-up outpatient care. SafeTy and Recovery Therapy (START) is a 4-session cognitive behavioral intervention augmented by mobile technology, which delivers automated and personalized reinforcement of adaptive coping behavior outside of the clinic setting. START builds from collaborative development alongside a community psychiatric service organization, and our preliminary data in the SMI population that supports the feasibility, acceptability, and impact of brief, mobile augmented cognitive behavioral intervention.

In a 3-year developmental study, our deployment focused approach will first refine intervention procedures, safety and care continuity protocols, and fit with the deployment setting with a series of collaborative contacts with community providers, project staff, advisors, and patient advocates. We will next conduct a pilot randomized controlled trial with 70 patients diagnosed with either bipolar disorder or schizophrenia rapidly referred by community triage providers to receive START in the walk-in clinic setting. Patients are enrolled who have SMI diagnoses and current active suicidal ideation and/or a suicide attempt in the prior 3 months. Participants are randomized to one of two active conditions: START + Mobile augmentation or START alone. We will evaluate feasibility, acceptability, and enhancement of rates of outpatient treatment engagement and crisis service use in comparison to the sample population. We will also examine pragmatic mechanisms, which include outpatient treatment engagement and coping self-efficacy, on change in suicidal ideation severity and crisis service use along with the preliminary impact of mobile augmentation.

ELIGIBILITY:
All subjects are recruited from San Diego area "walk-in" behavioral health evaluation services and must be referred by a triage clinician at such facilities. The study is unable to accept referrals from other sources. In addition, the following criteria apply:

Inclusion Criteria:

1. Subjects must have present suicidal ideation CSSR-S> 2 ("Active thoughts of killing oneself") in past 1 month and/or a suicide attempt in the prior 3 months as identified by the Columbia Suicide Severity Rating Scale
2. Diagnosis of DSM-V bipolar disorder, schizophrenia, or schizoaffective disorder as identified by the MINI International Neuropsychiatric Interview
3. Plans to remain in San Diego region for at least 6 months,
4. Capable of informed consent.

Exclusion Criteria:

1. Not English speaking
2. Cannot complete the assessment battery;
3. Insufficient visual acuity/manual dexterity for navigating a touch screen;
4. Current intoxication or substance use requiring immediate detoxification or outpatient plan directed at substance abuse services (versus mental health services which are separate in San Diego county);
5. Under conservatorship requiring proxy consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Scale for Suicide Ideation | Change in severity of suicide ideation over 24 weeks
  21 Item clinician rated scale

SECONDARY OUTCOMES:
Columbia Suicide Severity Rating Scale - Interval Version | Rate of suicidal behavior over 24 weeks
  Measure of the presence and severity of ideation and behavior over a defined interval

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parrish EM, Quynh A, Scott V, Chalker SA, Chang C, Kamarsu S, Twamley EW, Depp CA. Suicide Safety Plan Self-knowledge in Serious Mental Illness: Psychiatric Symptom Correlates and Effects of Brief Intervention. Community Ment Health J. 2023 Nov;59(8):1639-1646. doi: 10.1007/s10597-023-01155-5. Epub 2023 Jun 20. PMID 37340170
- [Derived] Depp CA, Parrish EM, Chalker SA, Ehret BC, Kamarsu S, Perivoliotis D, Granholm E. Pilot feasibility trial of a brief mobile-augmented suicide prevention intervention for serious mental illness. Psychiatr Rehabil J. 2023 Mar;46(1):74-82. doi: 10.1037/prj0000547. PMID 36809018
- [Derived] Depp C, Ehret B, Villa J, Perivoliotis D, Granholm E. A Brief Mobile-Augmented Suicide Prevention Intervention for People With Psychotic Disorders in Transition From Acute to Ongoing Care: Protocol for a Pilot Trial. JMIR Res Protoc. 2021 Feb 8;10(2):e14378. doi: 10.2196/14378. PMID 33555265